CLINICAL TRIAL: NCT03671044
Title: A Global, Multicenter, Three Arms, Open-label Randomized Study to Evaluate the Efficacy and Safety of Nanosomal Docetaxel Lipid Suspension Compared to Taxotere® (Docetaxel Injection Concentrate) in Triple-negative Breast Cancer Patients With Locally Advanced or Metastatic Breast Cancer After Failure to Prior Chemotherapy
Brief Title: A Study to Evaluate the Efficacy and Safety of Nanosomal Docetaxel Lipid Suspension in Triple Negative Breast Cancer Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jina Pharmaceuticals Inc. (Industry)
Collaborators: Intas Pharmaceuticals, Ltd. (Industry); Lambda Therapeutic Research Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0063-17
Record Dates: First submitted 2018-08-03; First posted 2018-09-14 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Triple Negative Breast Cancer
Keywords: Triple Negative Breast Cancer; Docetaxel
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Intervention Model Description: Experimental: T1, Nanosomal Docetaxel Lipid Suspension (75 mg/m2) Experimental: NDLS for Injection, 75 mg/ m2 Nanosomal Docetaxel Lipid Suspension for Injection; Dose: 75 mg/m2; Frequency: Every 3-weeks; Duration of treatment: Patient will be dosed with drug until disease progression and/or unacceptable toxicity.
  Experimental: T2, Nanosomal Docetaxel Lipid Suspension (100 mg/m2) Experimental: NDLS for Injection, 100 mg/ m2 Nanosomal Docetaxel Lipid Suspension for Injection; Dose: 100 mg/m2; Frequency: Every 3-weeks; Duration of treatment: Patient will be dosed with drug until disease progression and/or unacceptable toxicity.
  Active Comparator: R, Taxotere® (100 mg/m2) Active Comparator: Taxotere® Injection Concentrate Docetaxel Injection Concentrate; Dose: 100 mg/m2; Frequency: Every 3-weeks; Duration of treatment: Patient will be dosed with drug until disease progression and/or unacceptable toxicity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Nanosomal Docetaxel Lipid Suspension - 75 mg/m2 (Experimental): Experimental: NDLS for Injection, 75 mg/ m2 Nanosomal Docetaxel Lipid Suspension for Injection; Dose: 75 mg/m2; Frequency: Every 3-weeks; Duration of treatment: Patient will be dosed with drug until disease progression and/or unacceptable toxicity
  Interventions: Drug: Nanosomal Docetaxel Lipid Suspension (75 mg/m2)
- T2, Nanosomal Docetaxel Lipid Suspension (100 mg/m2) (Experimental): Experimental: NDLS for Injection, 100 mg/ m2 Nanosomal Docetaxel Lipid Suspension for Injection; Dose: 100 mg/m2; Frequency: Every 3-weeks; Duration of treatment: Patient will be dosed with drug until disease progression and/or unacceptable toxicity
  Interventions: Drug: Nanosomal Docetaxel Lipid Suspension (100 mg/m2)
- R, Taxotere® (100 mg/m2) (Active Comparator): Active Comparator: Taxotere® Injection Concentrate Docetaxel Injection Concentrate; Dose: 100 mg/m2; Frequency: Every 3-weeks; Duration of treatment: Patient will be dosed with drug until disease progression and/or unacceptable toxicity
  Interventions: Drug: Taxotere® (100 mg/m2)

INTERVENTIONS:
Drug: Nanosomal Docetaxel Lipid Suspension (75 mg/m2) — Each vial containing lyophilized Docetaxel lipid powder, equivalent to 20 mg or 80 mg of anhydrous Docetaxel.
  Arms: Nanosomal Docetaxel Lipid Suspension - 75 mg/m2
Drug: Nanosomal Docetaxel Lipid Suspension (100 mg/m2) — Each vial containing lyophilized Docetaxel lipid powder, equivalent to 20 mg or 80 mg of anhydrous Docetaxel.
  Arms: T2, Nanosomal Docetaxel Lipid Suspension (100 mg/m2)
Drug: Taxotere® (100 mg/m2) — Docetaxel Injection Concentrate; 20 mg/0.5 mL
  Arms: R, Taxotere® (100 mg/m2)

SUMMARY:
The Nanosomal Docetaxel Lipid Suspension (NDLS) consists of uniformly sized micro particles of docetaxel suspended in a lipid based formulation. The advantage of such a Lipid Based formulation of Docetaxel is an improvement of the safety profile by eliminating excipients, polysorbate 80 and ethanol which are present in conventional Docetaxel formulations (Taxotere®). This randomized, open-label study is designed to assess the efficacy and safety of Nanosomal Docetaxel Lipid Suspension at the dose of 75 mg/m2 and at the dose of 100 mg/m2 compared to Taxotere® at the dose of 100 mg/m2 in triple-negative breast cancer patients with Locally Advanced or Metastatic Breast Cancer. Patients will continue the treatment in the absence of disease progression and unacceptable toxicity. Disease status and tumor response will be assessed using Response Evaluation Criteria in Solid Tumors (RECIST 1.1) guidelines. 657 patients (219 patients per arm) will be randomized in the study. The trial will be conducted as per the ICH GCP Guidelines E6 (R1), Schedule Y (Amended Version 2013), Declaration of Helsinki (Fortaleza, Brazil, October 2013), ICMR Guidelines for Biomedical Research on Human subjects and in accordance with other applicable guidelines.

DETAILED DESCRIPTION:
Docetaxel is an antineoplastic agent belonging to the taxoid family. It is prepared by semi synthesis beginning with a precursor extracted from the renewable needle biomass of yew plants. It acts by disrupting the microtubular network in cells that is essential for mitotic and interphase cellular functions. The Nanosomal Docetaxel Lipid Suspension (NDLS) consists of uniformly sized micro particles of docetaxel suspended in a lipid based formulation. Docetaxel Lipid Suspension for Injection 20 mg/80 mg was approved for marketing in India. Intas Pharmaceuticals Ltd., is marketing this drug in India under the Brand name of DOCEAQUALIP 20/80 (Nanosomal Docetaxel Lipid Suspension for Injection 20/80 mg/vial) since 2013. This randomized, open label study is designed to assess the efficacy and safety of Nanosomal Docetaxel Lipid Suspension at the dose of 75 mg/m2 and at the dose of 100 mg/m2 compared to reference product, Taxotere® at a dose of 100 mg/m2 in triple-negative breast cancer patients with Locally Advanced or Metastatic Breast Cancer. 657 patients (219 patients per arm) will be randomized in the study.

To ensure consistent interpretation of measurable disease and objective endpoints for the study, all imaging studies performed throughout the study will be sent to an independent Central Radiological Facility for tumor measurement and evaluation of response. This independent review will have no impact on patient care. Continued participation in the study will be determined by assessment of clinical and radiological response by the Principal Investigator, and/or Radiologist. Efficacy evaluation will be done by CT scan/MRI and Bone scan at the end of treatment cycle 3 and will continue at every 3 cycles while the patient remains on treatment and compared to base line. Patient will continue study treatment until unacceptable toxicity or progression of disease. Patient will be screened up to 14 days prior to dosing and will be dosed on day 1. Patient will be advised to come in the facility at least 02 hours prior to dosing and will remain in the clinical facility until the completion of study drug administration. Dosing of patients will be done on ambulatory basis; hence patient hospitalization is optional. It is the responsibility of the PI to ensure that adequate medical supervision and care is available for the study patients during housing and entire duration of the study for utmost safety and wellbeing of the study patients. All safety analyses will be performed on the Safety set. Safety variables include AEs, clinical laboratory parameters, vital signs, physical examinations and electrocardiogram etc. Safety variables will be listed and summarized with descriptive statistics, as appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. The patient willing to give written signed and dated informed consent to participate in the study.
2. Patient must have histopathologically or cytologically confirmed triple negative breast cancer.
3. Patients may have received one prior chemotherapy regimen for adjuvant therapy and/or one chemotherapy treatment/regimen for firstline metastatic therapy
4. Patients with locally advanced or metastatic breast cancer after failure of prior chemotherapy.
5. Have at least one measurable lesion as per the RECIST criteria (version 1.1).
6. Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to two
7. Left Ventricular Ejection fraction (LVEF) greater than or equal to 50 percentage as per Echocardiography (ECHO).
8. Patient must have recovered from any toxic effects of previous chemotherapy or radiotherapy as judged by the Investigator.
9. Previous chemotherapy or radiotherapy should be completed 4 weeks prior to start of IMP administration.
10. Patients with life expectancy of at least 6 months.
11. Serum pregnancy test at screening and urine pregnancy test on Day 1 (before randomization) must be negative.
12. Sexually active women, unless surgically sterile or postmenopausal for at least 12 consecutive months, must use an effective method of avoiding pregnancy (including oral, transdermal, or implanted contraceptives [any hormonal method in conjunction with a secondary method], intrauterine device, female condom with spermicide, diaphragm with spermicide, absolute sexual abstinence, use of condom with spermicide by sexual partner or sterile [at least 6 months prior to Study drug administration] sexual partner) for at least four weeks prior to study drug administration, during study and up to 30 days after the last dose of study drug. Cessation of birth control after this point should be discussed with a responsible physician.
13. Patient with adequate bone marrow, renal and hepatic function.

Exclusion Criteria:

1. Patient who has a history of hypersensitivity reactions to Docetaxel or any other component of formulation or to any drugs formulated with polysorbate 80.
2. Patients with a history of HER2 positive over expression and hormone receptor positive (ER or PR)
3. Patient who is already exposed to Docetaxel injection in metastatic setting.
4. Any of the cardiac conditions like Unstable angina, Myocardial infarction within the past six months, Severe uncontrolled ventricular arrhythmias, Clinically significant pericardial disease, Electrocardiographic evidence of acute ischemia, Patient with evidence of abnormal cardiac conduction (e.g., bundle branch block or heart block) except in whom the disease has been stable for the past six months, History of cardiac disease that met the NYHA Classification class 2 or greater
5. Uncontrolled diabetes or infection.
6. Known history of drug addiction within last one year.
7. Patients with known CNS lesions (brain metastasis or carcinomatous meningitis) except for asymptomatic brain metastases.
8. The receipt of an investigational medicinal product or participation in other drug research study within a period of 30 days prior to the first dose of investigational medicinal Product for the current study.
9. Pre-existing motor or sensory neurotoxicity of a severity greater than or equal to grade two as defined by NCI CTCAE 4.03 criteria.
10. Known case of HIV infection.
11. Any other condition that, in the investigator's judgment, might increase the risk to the patient or decrease the chance of obtaining satisfactory data needed to achieve the objectives of the study.
12. Patients who are unwilling or unable to follow protocol requirements

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 657 (Estimated)
Dates: Start 2018-07-10 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of the patients with Objective Response Rate (i.e., CR + PR) as the Best Overall Response Rate (i.e., CR + PR) in the test arm (NDLS) compared to reference arm (Taxotere) | Approximately 2 years after study initiation
  Non-inferiority of NDLS (75 mg/m2, 100 mg/m2) compared to Taxotere (100 mg/m2)

SECONDARY OUTCOMES:
Progression free survival (PFS) | Approximately 2 years after study initiation
  PFS will be evaluated from the date of first dosing to the date of tumor progression (as per the RECIST 1.1 Criteria) or death (due to any cause) whichever occurred first
To evaluate the overall survival (OS) of the patients | Approximately 2 years after study initiation
  OS will be evaluated from the date of first dosing to the date of tumor progression (as per the RECIST 1.1 Criteria) or death (due to any cause) whichever occurred first
Incidence of adverse events as assessed by clinical examination, and/or laboratory parameters | Approximately 2 years after study initiation
  adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ravi Alamchandani, Study Chair — Lambda Therapeutic Research Ltd.
Locations (4):
- United States (3):
  - Columbus Regional Research Institute, LLC, Columbus, Georgia
  - Cox Medical Center, Springfield, Missouri
  - Gabrail Cancer Center, Canton, Ohio
- Kailash Cancer Hospital & Research Centre, Vadodara, Gujarat, India

REFERENCES:
- [Derived] Subramanian S, Prasanna R, Biswas G, Das Majumdar SK, Joshi N, Bunger D, Khan MA, Ahmad I. Nanosomal Docetaxel Lipid Suspension-Based Chemotherapy in Breast Cancer: Results from a Multicenter Retrospective Study. Breast Cancer (Dove Med Press). 2020 May 22;12:77-85. doi: 10.2147/BCTT.S236108. eCollection 2020. PMID 32547188